CLINICAL TRIAL: NCT00924014
Title: Comparative Effects of Conivaptan and Loop Diuretics on Plasma Neurohormones and Systemic and Renal Hemodynamics in Subjects With Chronic Congestive Heart Failure
Brief Title: Comparing the Effects of Conivaptan and Diuretics on Plasma Neurohormones and Renal Blood Flow in Patients With Chronic Congestive Heart Failure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hennepin County Medical Center, Minneapolis (Other)
Collaborators: Astellas Pharma Inc (Industry)
Responsible Party: Steven R. Goldsmith, Hennepin County Medical Center
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 001; IND 104, 334
Record Dates: First submitted 2009-06-17; First posted 2009-06-18 (Estimated); Last update posted 2009-06-18 (Estimated); Status verified 2009-06

CONDITIONS: Heart Failure
Keywords: heart failure
MeSH Terms: conditions — Heart Failure | interventions — conivaptan; Furosemide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Conivaptan (Active Comparator): Conivaptan will be given via IV bolus
  Interventions: Drug: Conivaptan
- Furosemide (Active Comparator): Furosemide will be given via IV bolus
  Interventions: Drug: Furosemide
- conivaptan and furosemide (Active Comparator): on day 3 subjects will receive both study drugs
  Interventions: Drug: Conivaptan and furosemide

INTERVENTIONS:
Drug: Conivaptan — Conivaptan 20 mg IV bolus followed by a 4 hour infusion at 1.2 mg/hr
  Other Names: vaprisol
  Arms: Conivaptan
Drug: Furosemide — Furosemide will be given IV at the subjects usual oral dose up to 80 mg. If the dose is 80 mg or more only 1/2 the dose will be given IV.
  Other Names: Lasix
  Arms: Furosemide
Drug: Conivaptan and furosemide — Furosemide bolus first; conivaptan 20 mg IV bolus/infusion at 1.2 mg/hour for a total of 4 hours
  Other Names: vaprisol; lasix
  Arms: conivaptan and furosemide

SUMMARY:
The purpose of the study is to compare the effects of conivaptan and diuretics on renal blood flow and neurohormones.

DETAILED DESCRIPTION:
1. To define the hemodynamic, neurohormonal and renal responses to intravenous conivaptan in patients with chronic stable heart failure (HF), and compare these responses to those after intravenous furosemide.
2. To define the hemodynamic, neurohormonal and renal responses to the combination of the two drugs (conivaptan and furosemide).

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of chronic congestive heart failure of any etiology
* Be between 18-80 years of age
* Able to provide consent
* Have a documented left ventricular ejection fraction within the last year of < 40%
* On a stable dose (no changes within 2 weeks) of 40 mg or greater daily dose of furosemide or its equivalent
* On standard HF therapy medications (ACEI or ARB and beta-blocker unless contraindicated)
* Have an estimated glomerular filtration rate (GFR) of 30 ml/minute or greater (based on the Cockcroft Gault calculation)
* Have a hemoglobin of > 10 grams/dl
* Have a negative urine pregnancy for women of childbearing years only

Exclusion Criteria:

* Acute coronary syndrome within 1 month
* Systolic blood pressure less than or equal to 90 mmHg at time of enrollment
* Poor peripheral venous access
* Severe concomitant disease which deemed by the investigator would render them unsuitable for this trial
* Allergy or contraindication to the use of iothalamate, PAH - Specifically any allergies to iodine or iodine containing products, history of asthma and hay fever which deemed by the investigator would render them unsuitable for this trial

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2009-07; Primary Completion 2009-12 (Estimated); Study Completion 2010-03 (Estimated)

PRIMARY OUTCOMES:
renal hemodynamics renal blood flow and glomerular filtration rate | measured on days 1, 2, 3

SECONDARY OUTCOMES:
measure plasma neurohormone levels | predose, 1 hour and 4 hours post dose measured on day 1, 2, 3

CONTACTS AND LOCATIONS:
Overall Officials: Steven R Goldsmith, MD, Study Director — Hennepin County Medical Center, Minneapolis
Locations (1):
- Hennepin county Medical Center, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Goldsmith SR, Gilbertson DT, Mackedanz SA, Swan SK. Renal effects of conivaptan, furosemide, and the combination in patients with chronic heart failure. J Card Fail. 2011 Dec;17(12):982-9. doi: 10.1016/j.cardfail.2011.08.012. Epub 2011 Oct 6. PMID 22123359